CLINICAL TRIAL: NCT04506905
Title: A 2-Part Randomized Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Alternate MK-8189 Titration Regimens in Young Adult Participants With Schizophrenia and to Evaluate the Safety, Tolerability and Pharmacokinetics of MK-8189 in Elderly Participants With Schizophrenia and Healthy Elderly
Brief Title: Safety, Tolerability, and Pharmacokinetics Study of MK-8189 in Participants With Schizophrenia and Healthy Participants (MK-8189-011)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8189-011; Merck Protocol Number (Other: MK-8189-011)
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — MK-8189

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part 1 (Panel A) MK-8189 (Experimental): Young adult participants with schizophrenia receive MK-8189 titrated from 16 mg to 24 mg once daily (QD), orally, over a course of 7-day treatment.
  Interventions: Drug: MK-8189
- Part 1 (Panel B) MK-8189 (Experimental): Young adult participants with schizophrenia receive MK-8189 titrated up to 24 mg QD, orally, over a course of 7-day treatment period with starting doses based on safety and tolerability of previous starting dose in previous panel.
  Interventions: Drug: MK-8189
- Part 1 (Panel C) MK-8189 (Experimental): Young adult participants with schizophrenia receive MK-8189 titrated from 8 mg to 24 mg QD, orally, over a course of 7-day treatment period with starting doses based on safety and tolerability of previous starting dose in previous panels.
  Interventions: Drug: MK-8189
- Part 2 (Panel D) MK-8189 (Experimental): Elderly adult participants with schizophrenia receive MK-8189 titrated from 8 mg to 24 mg QD, orally, over the course of a 13-day treatment period with starting doses based on safety and tolerability of previous starting dose in previous panels.
  Interventions: Drug: MK-8189
- Part 2 (Panel E) MK-8189 (Experimental): Elderly adult participants with schizophrenia receive MK-8189 titrated from 16 mg to 24 mg QD, orally, over the course of 10-day treatment period with starting doses based on safety and tolerability of previous starting dose in previous panels.
  Interventions: Drug: MK-8189
- Part 2 (Panel F) MK-8189 (Experimental): Healthy elderly adult participants receive MK-8189 titrated from 8 mg to 24 mg QD, orally, over the course of a 13-day treatment period with starting doses based on safety and tolerability of previous starting dose in previous panels.
  Interventions: Drug: MK-8189
- Part 2 (Panel G) MK-8189 (Experimental): Healthy elderly adult participants receive MK-8189 titrated from 16 mg to 24 mg QD, orally, over the course of 10-day treatment period with starting doses based on safety and tolerability of previous starting dose in previous panels.
  Interventions: Drug: MK-8189
- Part 1 (Panels A, B, C) Placebo (Placebo Comparator): Oral tablets of dose-matched placebo to total daily dose of MK-8189.
  Interventions: Drug: Placebo
- Part 2 (Panels D, E, F, G) Placebo (Placebo Comparator): Oral tablets of dose-matched placebo to total daily dose of MK-8189.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8189 — MK-8189, oral, 4 mg and/or 12 mg tablets for a total daily dose of 8, 16 or 24 mg QD according to randomization
  Arms: Part 1 (Panel A) MK-8189; Part 1 (Panel B) MK-8189; Part 1 (Panel C) MK-8189; Part 2 (Panel D) MK-8189; Part 2 (Panel E) MK-8189; Part 2 (Panel F) MK-8189; Part 2 (Panel G) MK-8189
Drug: Placebo — Oral tablets of dose-matched placebo to MK-8189 according to randomization
  Arms: Part 1 (Panels A, B, C) Placebo; Part 2 (Panels D, E, F, G) Placebo

SUMMARY:
This is a randomized, double-blind, 2-part clinical study of the safety, tolerability and pharmacokinetics of alternate MK-8189 titration regimens. Part 1 assessed multiple dose once-daily titration regimens of MK-8189 in young adult participants with schizophrenia. Part 2 assessed multiple once-daily doses of MK-8189 in elderly participants with schizophrenia and healthy elderly participants.

ELIGIBILITY:
Inclusion Criteria:

* Has a body mass index (BMI) ≤40 kg/m2
* Has no clinically significant abnormality on 12-lead safety electrocardiogram (ECG) performed at the prestudy (screening) visit and/or prior to randomization
* Has a normal resting blood pressure (BP: systolic BP is ≥90 millimeter of mercury [mmHg] and ≤140 mmHg; diastolic BP is ≥60 mmHg and ≤90 mmHg) and normal resting heart rate (≥45 beats per minute [bpm] and ≤100 bpm) in the semirecumbent position at the prestudy (screening) visit and/or prior to randomization. Repeat evaluations may be done if the values for a participant are, per investigator discretion, minimally outside the designated range. Participants may be included if values are outside the normal range but considered not clinically significant per investigator discretion
* Participants with schizophrenia only: Meets diagnostic criteria for schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria with the onset of the first episode being no less than 2 years prior to screening and monotherapy with antipsychotics for treatment should be indicated
* Participants with schizophrenia only: Has a total Brief Psychiatric Rating Scale (BPRS) score of <48 with a BPRS score <4 for #10 (hostility) and #14 (uncooperativeness) at the screening visit
* Participants with schizophrenia only: Is in the nonacute phase of their illness and clinically stable for 3 months prior to screening as demonstrated by the following: 1) no clinically significant change in dose of prescribed antipsychotic medication, or clinically significant change in antipsychotic medication to treat symptoms of schizophrenia for 2 months prior to screening 2) no increase in level of psychiatric care due to worsening of symptoms of schizophrenia for 3 months prior to screening
* Participants with schizophrenia only: Has a history of receiving and tolerating antipsychotic medication within the usual dose range employed for schizophrenia
* Participants with schizophrenia only: Has a stable living situation
* Participants with hypothyroidism, diabetes, high BP, chronic respiratory conditions or other mild forms of these medical conditions could be considered as candidates for study enrollment if their condition is stable
* Has regular bowel movements
* Participants with schizophrenia only: Is able to discontinue the use of all antipsychotic medication at least 5 days prior to the start of the treatment period and during the study period
* Female participants are not pregnant and not breastfeeding, and are not a woman of childbearing potential (WOCBP) or are a WOCBP who agrees to follow contraceptive guidance during the treatment period and for at least 14 days after the last dose of study intervention

Exclusion Criteria:

* Is a WOCBP who has a positive urine pregnancy test within 48 hours before the first dose of study intervention
* Participants with schizophrenia only: Has evidence or history of a primary DSM-5 axis I psychiatric diagnosis other than schizophrenia or schizoaffective disorder per the allowed DSM-5 criteria within 1 month of screening
* Has evidence or history of a primary DSM-5 axis I psychiatric diagnosis other than schizophrenia or schizoaffective disorder per the allowed DSM-5 criteria within 1 month of screening
* Has evidence or history of mental retardation, borderline personality disorder, anxiety disorder, or organic brain syndrome
* Has a history of neuroleptic malignant syndrome or moderate to severe tardive dyskinesia
* Has a substance-induced psychotic disorder or behavioral disturbance thought to be due to substance abuse
* Has a DSM-5 defined substance use disorder within 3 months of screening
* Has a history of seizure disorder beyond childhood or is receiving treatment with any anticonvulsant to prevent seizures
* Has an untreated or uncompensated clinically significant renal, endocrine, hepatic, respiratory, gastrointestinal, psychiatric, neurologic, cardiovascular, hematological, immunological or cerebrovascular disease, malignancy, allergic disease or other chronic and/or degenerative process at screening
* Has any clinically significant abnormal laboratory, vital sign (VS), physical examination, or 12-lead safety ECG findings at screening or changes from baseline parameters or, in the opinion of the investigator, would make the participant inappropriate for entry into this study
* Has a history of cancer with following exceptions: 1) Adequately treated nonmelanomatous skin carcinoma or carcinoma in situ of the cervix or; 2) Other malignancies which have been successfully treated with appropriate follow up and therefore unlikely to recur for the duration of the study, in the opinion of the investigator and with agreement of the Sponsor
* Has a clinically significant history or presence of sick sinus syndrome, first, second, or third-degree AV block, myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged corrected QT (QTc) interval, or conduction abnormalities
* Has history of repeated or frequent syncope, vasovagal episodes, or epileptic seizures
* Has a family history of sudden death
* Has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the participant by their participation in the study
* For Part 2 participants only: Participant has an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 based on the modification of diet in renal disease (MDRD). Participants who have an eGFR or measured creatinine clearance of up to10% below of either 60 milliliter/minute [mL/min] (for creatinine clearance) or 60 mL/min/1.73m2 (for eGFR) may be enrolled in the study at the discretion of the investigator
* Has a history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Is positive for Hepatitis B surface antigen, Hepatitis C antibodies or HIV
* Had major surgery, donated or lost 1 unit of blood within 4 weeks prior to the prestudy (screening) visit
* Healthy participants only: Is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years (participants who have had situational depression may be enrolled in the study at investigator's discretion)
* Participants with schizophrenia only: Is at imminent risk of self-harm, based on clinical interview and responses on the Columbia-Suicide Severity Rating Scale (C-SSRS), or of harm to others in the opinion of the investigator
* Healthy participants only: Is at imminent risk of self-harm, based on clinical interview and responses on the CSSRS, or of harm to others in the opinion of the investigator. Participants must be excluded if they report suicidal ideation with intent, with or without a plan or in the past 5 years or suicidal behavior in their lifetime
* Has received treatment with clozapine for schizophrenia or treatment with monoamine oxidase inhibitors within 3 months of screening or cariprazine within 2 months of screening
* Has received a parenteral depot antipsychotic medication within 3 months of screening
* Is unable to refrain from the use of co-medication with a moderate or strong inhibiting or inducing effect on cytochrome (CYP3A) and/or cytochrome (CYP2C9) beginning approximately 2 weeks or 5 half-lives, whichever is longer, prior to administration of the initial dose of trial drug and throughout the trial or is unable to refrain from the use of sensitive substrates of cytochrome (CYP2B6)
* Has participated in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to the prestudy (screening) visit
* Has been in incarceration or imprisonment within three months prior to screening
* Is a current smoker (healthy participants only) or is a smoker (participants with schizophrenia only) that does not agree to follow the smoking restrictions as defined by the clinical research unit (CRU)
* Consumes greater than 3 glasses of alcoholic beverages per day. Participants who consume 4 glasses of alcoholic beverages per day may be enrolled at the discretion of the investigator
* Consumes excessive amounts, defined as greater than 6 servings of caffeinated beverages per day
* Is a regular user of cannabis, any illicit drugs or has a history of drug abuse within approximately 3 years
* Presents any concern by the investigator regarding safe participation in the study or for any other reason the investigator considers the participant inappropriate for participation in the study
* Is or has an immediate family member who is investigational site or Sponsor staff directly involved with this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (6):
- United States (6):
  - Woodland Research Northwest, LLC ( Site 0002), Rogers, Arkansas
  - Parexel ( Site 0004), Glendale, California
  - Collaborative NeuroScience Network ( Site 0008), Long Beach, California
  - Velocity Clinical Research, Hallandale Beach ( Site 0001), Hallandale, Florida
  - RCA at Fort Lauderdale Behavioral Health Center ( Site 0006), Oakland Park, Florida
  - Hassman Research Institute ( Site 0007), Berlin, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 6 study centers in USA.
Groups:
- Part 1, Panel A: MK-8189 16 mg to 24 mg: Young adult participants with schizophrenia receive MK-8189 titrated from 16 mg (Days 1 to 3) to 24 mg (Days 4 to 7) QD for 7 days.
- Part 1, Panel B: MK-8189 24 mg: Young adult participants with schizophrenia receive MK-8189 24 mg QD from Day 1 to Day 7.
- Part 1, Panel C: MK-8189 8 mg t0 24 mg: Young adult participants with schizophrenia were planned to receive MK-8189 titrated from 8 mg to 24 mg QD over 7 days.
- Part 2, Panel D: MK-8189 8 mg to 24 mg: Elderly adult participants with schizophrenia receive MK-8189 titrated from 8 mg (Days 1 to 3), to 16 mg (Days 4 to 7), to 24 mg (Days 7 to 13) QD over 13 days.
- Part 2, Panel E: MK-8189 16 mg to 24 mg: Elderly adult participants with schizophrenia were intended to receive MK-8189 titrated from 16 mg to 24 mg QD, over 10 days.
- Part 2, Panel F: MK-8189 8 mg to 24 mg: Healthy elderly adult participants receive receive MK-8189 titrated from 8 mg (Days 1 to 3), to 16 mg (Days 4 to 7), to 24 mg (Days 7 to 13) QD over 13 days.
- Part 2, Panel G: MK-8189 16 mg to 24 mg: Healthy elderly adult participants receive MK-8189 titrated from 16 mg (Days 1 to 3), to 24 mg (Days 4 to 10) QD over 10 days.
- Part 1: Placebo: Young adult participants with schizophrenia receive placebo matched to MK-8189 QD for 7 days.
- Part 2: Placebo: Elderly participants with schizophrenia and heathy elderly participants receive placebo matched to MK-8189 for up to 13 days.
Period: Overall Study
Arm/Group | Part 1, Panel A: MK-8189 16 mg to 24 mg | Part 1, Panel B: MK-8189 24 mg | Part 1, Panel C: MK-8189 8 mg t0 24 mg | Part 2, Panel D: MK-8189 8 mg to 24 mg | Part 2, Panel E: MK-8189 16 mg to 24 mg | Part 2, Panel F: MK-8189 8 mg to 24 mg | Part 2, Panel G: MK-8189 16 mg to 24 mg | Part 1: Placebo | Part 2: Placebo
Started | 6 | 14 | 0 (Panel C was never initiated.) | 12 | 0 (Panel E was never initiated.) | 5 | 13 | 6 | 7
Completed | 5 | 14 | 0 | 9 | 0 | 5 | 13 | 6 | 7
Not Completed | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrollment into Part 1 Panel C, and Part 2 Panel E, was never initiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, Panel A: MK-8189 16 mg to 24 mg | Part 1, Panel B: MK-8189 24 mg | Part 1, Panel C: MK-8189 8 mg t0 24 mg | Part 2, Panel D: MK-8189 8 mg to 24 mg | Part 2, Panel E: MK-8189 16 mg to 24 mg | Part 2, Panel F: MK-8189 8 mg to 24 mg | Part 2, Panel G: MK-8189 16 mg to 24 mg | Part 1: Placebo | Part 2: Placebo | Total
Number analyzed (Participants) | 6 | 14 | 0 | 12 | 0 | 5 | 13 | 6 | 7 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (8.8) | 44.9 (10.8) |  | 64.2 (2.0) |  | 69.4 (2.3) | 68.4 (3.6) | 43.3 (8.6) | 66.3 (4.7) | 57.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 5 | 0 | 1 | 10 | 1 | 5 | 25
  Male | 5 | 12 | 0 | 7 | 0 | 4 | 3 | 5 | 2 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 0 | 0 | 3 | 9 | 0 | 3 | 18
  Not Hispanic or Latino | 4 | 13 | 0 | 11 | 0 | 2 | 4 | 6 | 4 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 11 | 0 | 9 | 0 | 0 | 2 | 5 | 4 | 34
  White | 3 | 2 | 0 | 2 | 0 | 5 | 11 | 1 | 3 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1 & 2: Number of Participants Who Experienced an Adverse Event (AE)
Description: The number of participants with ≥1 AE is reported. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to approximately 27 days
Population: All randomized and treated participants are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1, Panel A: MK-8189 16 mg to 24 mg | Part 1, Panel B: MK-8189 24 mg | Part 1, Panel C: MK-8189 8 mg t0 24 mg | Part 2, Panel D: MK-8189 8 mg to 24 mg | Part 2, Panel E: MK-8189 16 mg to 24 mg | Part 2, Panel F: MK-8189 8 mg to 24 mg | Part 2, Panel G: MK-8189 16 mg to 24 mg | Part 1: Placebo | Part 2: Placebo
Number analyzed (Participants) | 6 | 14 | 0 | 12 | 0 | 5 | 13 | 6 | 7
Participants | 4 | 9 |  | 3 |  | 2 | 8 | 2 | 4

2. Primary Outcome: Part 1 & 2: Number of Participants Discontinuing Study Treatment Due to an AE
Description: The number of participants discontinuing from study treatment due to ≥1 AE is reported. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Time Frame: Up to approximately 27 days
Population: All randomized and treated participants are included.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1, Panel B: MK-8189 24 mg: Young adult participants with schizophrenia receive MK-8189 24 mg QD for 7 days.
Arm/Group | Part 1, Panel A: MK-8189 16 mg to 24 mg | Part 1, Panel B: MK-8189 24 mg | Part 1, Panel C: MK-8189 8 mg t0 24 mg | Part 2, Panel D: MK-8189 8 mg to 24 mg | Part 2, Panel E: MK-8189 16 mg to 24 mg | Part 2, Panel F: MK-8189 8 mg to 24 mg | Part 2, Panel G: MK-8189 16 mg to 24 mg | Part 1: Placebo | Part 2: Placebo
Number analyzed (Participants) | 6 | 14 | 0 | 12 | 0 | 5 | 13 | 6 | 7
Participants | 0 | 1 |  | 2 |  | 1 | 3 | 0 | 1

3. Secondary Outcome: Part 1: Area Under the Concentration Time-curve From Hour 0 to 24 Hours Postdose (AUC0-24) of MK-8189
Description: AUC0-24 was determined for participants in Part 1 panels who received MK-8189.
Time Frame: Days 1, 2, 4, and Day 7: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: Part 1 participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Least Squares Mean (95% Confidence Interval); unit: hr*nmol/L
Groups:
- Part 1, Panel A: MK-8189 16 mg: The PK of MK-8189 16 mg was assessed on Day 1 in Panel A.
- Part 1, Panel A: MK-8189 24 mg Day 4: The PK of MK-8189 24 mg was assessed on Day 4 in Panel A.
- Part 1, Panel A: MK-8189 24 mg Day 7: The PK of MK-8189 24 mg was assessed on Day 7 in Panel A.
- Part 1, Panel B: MK-8189 24 mg Day 1: The PK of MK-8189 24 mg was assessed on Day 1 in Panel B.
- Part 1, Panel B: MK-8189 24 mg Day 2: The PK of MK-8189 24 mg was assessed on Day 2 in Panel B.
- Part 1, Panel B: MK-8189 24 mg Day 7: The PK of MK-8189 24 mg was assessed on Day 7 in Panel B.
Arm/Group | Part 1, Panel A: MK-8189 16 mg | Part 1, Panel A: MK-8189 24 mg Day 4 | Part 1, Panel A: MK-8189 24 mg Day 7 | Part 1, Panel B: MK-8189 24 mg Day 1 | Part 1, Panel B: MK-8189 24 mg Day 2 | Part 1, Panel B: MK-8189 24 mg Day 7
Number analyzed (Participants) | 6 | 5 | 5 | 14 | 13 | 10
hr*nmol/L | 10500 [6210 to 17600] | 21200 [12600 to 35800] | 22700 [13500 to 38300] | 12500 [9920 to 15900] | 17600 [13800 to 22300] | 20500 [16000 to 26300]

4. Secondary Outcome: Part 1: Concentration 24 Hours Postdose (C24) of MK-8189
Description: C24 was determined for participants in Part 1 panels who received MK-8189.
Time Frame: Days 1, 2, 4, and Day 7: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Part 1, Panel A: MK-8189 16 mg | Part 1, Panel A: MK-8189 24 mg Day 4 | Part 1, Panel A: MK-8189 24 mg Day 7 | Part 1, Panel B: MK-8189 24 mg Day 1 | Part 1, Panel B: MK-8189 24 mg Day 2 | Part 1, Panel B: MK-8189 24 mg Day 7
Number analyzed (Participants) | 6 | 5 | 5 | 14 | 13 | 10
nmol/L | 615 [225 to 1680] | 322 [107 to 968] | 669 [223 to 2010] | 565 [389 to 821] | 567 [387 to 830] | 666 [445 to 997]

5. Secondary Outcome: Part 1: Maximum Plasma Concentration (Cmax) of MK-8189
Description: Cmax was determined for participants in Part 1 panels who received MK-8189.
Time Frame: Days 1, 2, 3, 4, and Day 7: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Groups:
- Part 1, Panel B: MK-8189 24 mg Day 3: The PK of MK-8189 24 mg was assessed on Day 3 in Panel B.
Arm/Group | Part 1, Panel A: MK-8189 16 mg | Part 1, Panel A: MK-8189 24 mg Day 4 | Part 1, Panel A: MK-8189 24 mg Day 7 | Part 1, Panel B: MK-8189 24 mg Day 1 | Part 1, Panel B: MK-8189 24 mg Day 2 | Part 1, Panel B: MK-8189 24 mg Day 3 | Part 1, Panel B: MK-8189 24 mg Day 7
Number analyzed (Participants) | 6 | 5 | 5 | 14 | 13 | 13 | 10
nmol/L | 700 [405 to 1210] | 1220 [707 to 2110] | 1270 [738 to 2200] | 941 [737 to 1200] | 996 [779 to 1270] | 956 [748 to 1220] | 1200 [933 to 1540]

6. Secondary Outcome: Part 1: Time to Maximum Concentration (Tmax) of MK-8189
Description: Tmax was determined for participants in Part 1 panels who received MK-8189.
Time Frame: Days 1, 2, 3, 4, and Day 7: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1, Panel A: MK-8189 16 mg | Part 1, Panel A: MK-8189 24 mg Day 4 | Part 1, Panel A: MK-8189 24 mg Day 7 | Part 1, Panel B: MK-8189 24 mg Day 1 | Part 1, Panel B: MK-8189 24 mg Day 2 | Part 1, Panel B: MK-8189 24 mg Day 3 | Part 1, Panel B: MK-8189 24 mg Day 7
Number analyzed (Participants) | 6 | 5 | 5 | 14 | 13 | 13 | 10
Hours | 19.97 [12.02 to 24.08] | 16.00 [10.00 to 23.97] | 16.00 [12.00 to 16.00] | 16.00 [2.00 to 23.97] | 8.00 [0.00 to 23.97] | 8.00 [0.00 to 8.00] | 11.03 [6.05 to 16.08]

7. Secondary Outcome: Part 1: Clearance (CL/F) of MK-8189
Description: CL/F was determined for participants in Part 1 panels who received MK-8189.
Time Frame: Day 7: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Part 1, Panel A: MK-8189 24 mg Day 7 | Part 1, Panel B: MK-8189 24 mg Day 7
Number analyzed (Participants) | 5 | 10
L/hr | 3.21 (36.5) | 3.22 (48.1)

8. Secondary Outcome: Part 1: Apparent Terminal Half-life (t½) of MK-8189
Description: t½ was determined for participants in Part 1 panels who received MK-8189.
Time Frame: Day 7: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1, Panel A: MK-8189 24 mg Day 7 | Part 1, Panel B: MK-8189 24 mg Day 7
Number analyzed (Participants) | 5 | 10
Hours | 7.99 (15.6) | 8.68 (26.8)

9. Secondary Outcome: Part 1: Volume of Distribution (Vd/F) of MK-8189
Description: Vd/F was determined for participants in Part 1 panels who received MK-8189.
Time Frame: Day 7: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1, Panel A: MK-8189 24 mg Day 7 | Part 1, Panel B: MK-8189 24 mg Day 7
Number analyzed (Participants) | 5 | 10
Liters | 37.03 (28.5) | 40.31 (40.4)

10. Secondary Outcome: Part 2: AUC0-24 of MK-8189
Description: AUC0-24 was determined for participants in Part 2 panels who received MK-8189.
Time Frame: Days 1, 4, 7, 10, and 13: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: Part 2 participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Least Squares Mean (95% Confidence Interval); unit: hr*nmol/L
Groups:
- Part 2, Panel D: MK-8189 8 mg: The PK of MK-8189 8 mg was assessed on Day 1 in Panel D.
- Part 2, Panel D: MK-8189 16 mg: The PK of MK-8189 16 mg was assessed on Day 4 in Panel D.
- Part 2, Panel D: MK-8189 24 mg: The PK of MK-8189 24 mg was assessed on Day 7 in Panel D.
- Part 2, Panel D: MK-8189 24 mg Day 13: The PK of MK-8189 24 mg was assessed on Day 13 in Panel D.
- Part 2, Panel F: MK-8189 8 mg: The PK of MK-8189 8 mg was assessed on Day 1 in Panel F.
- Part 2, Panel F: MK-8189 16 mg: The PK of MK-8189 16 mg was assessed on Day 4 in Panel F.
- Part 2, Panel F: MK-8189 24 mg: The PK of MK-8189 24 mg was assessed on Day 7 in Panel F.
- Part 2, Panel F: MK-8189 24 mg Day 13: The PK of MK-8189 24 mg was assessed on Day 13 in Panel F.
- Part 2, Panel G: MK-8189 16 mg: The PK of MK-8189 16 mg was assessed on Day 1 in Panel G.
- Part 2, Panel G: MK-8189 24 mg: The PK of MK-8189 24 mg was assessed on Day 4 in Panel G.
- Part 2, Panel G: MK-8189 24 mg Day 10: The PK of MK-8189 24 mg was assessed on Day 10 in Panel G.
Arm/Group | Part 2, Panel D: MK-8189 8 mg | Part 2, Panel D: MK-8189 16 mg | Part 2, Panel D: MK-8189 24 mg | Part 2, Panel D: MK-8189 24 mg Day 13 | Part 2, Panel F: MK-8189 8 mg | Part 2, Panel F: MK-8189 16 mg | Part 2, Panel F: MK-8189 24 mg | Part 2, Panel F: MK-8189 24 mg Day 13 | Part 2, Panel G: MK-8189 16 mg | Part 2, Panel G: MK-8189 24 mg | Part 2, Panel G: MK-8189 24 mg Day 10
Number analyzed (Participants) | 12 | 12 | 9 | 8 | 5 | 5 | 5 | 3 | 13 | 10 | 10
hr*nmol/L | 4600 [3210 to 6590] | 12400 [8620 to 17700] | 17100 [11400 to 25500] | 24000 [15800 to 36400] | 5930 [3800 to 9250] | 13800 [8820 to 21500] | 23600 [15100 to 36900] | 27800 [17800 to 43500] | 9860 [7810 to 12500] | 23500 [18300 to 30300] | 26800 [20600 to 34800]

11. Secondary Outcome: Part 2: C24 of MK-8189
Description: C24 was determined for participants in Part 2 panels who received MK-8189.
Time Frame: Days 1, 4, 7, 10, and 13: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Part 2, Panel D: MK-8189 8 mg | Part 2, Panel D: MK-8189 16 mg | Part 2, Panel D: MK-8189 24 mg | Part 2, Panel D: MK-8189 24 mg Day 13 | Part 2, Panel F: MK-8189 8 mg | Part 2, Panel F: MK-8189 16 mg | Part 2, Panel F: MK-8189 24 mg | Part 2, Panel F: MK-8189 24 mg Day 13 | Part 2, Panel G: MK-8189 16 mg | Part 2, Panel G: MK-8189 24 mg | Part 2, Panel G: MK-8189 24 mg Day 10
Number analyzed (Participants) | 12 | 12 | 9 | 8 | 5 | 5 | 5 | 3 | 13 | 11 | 10
nmol/L | 302 [187 to 488] | 508 [314 to 820] | 637 [370 to 1100] | 926 [522 to 1640] | 349 [212 to 575] | 612 [372 to 1010] | 927 [563 to 1530] | 1260 [721 to 2220] | 569 [409 to 790] | 885 [618 to 1270] | 1090 [748 to 1590]

12. Secondary Outcome: Part 2: Cmax of MK-8189
Description: Cmax was determined for participants in Part 2 panels who received MK-8189.
Time Frame: Days 1, 4, 7, 10, and 13: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: as for outcome 10
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Part 2, Panel D: MK-8189 8 mg | Part 2, Panel D: MK-8189 16 mg | Part 2, Panel D: MK-8189 24 mg | Part 2, Panel D: MK-8189 24 mg Day 13 | Part 2, Panel F: MK-8189 8 mg | Part 2, Panel F: MK-8189 16 mg | Part 2, Panel F: MK-8189 24 mg | Part 2, Panel F: MK-8189 24 mg Day 13 | Part 2, Panel G: MK-8189 16 mg | Part 2, Panel G: MK-8189 24 mg | Part 2, Panel G: MK-8189 24 mg Day 10
Number analyzed (Participants) | 12 | 12 | 9 | 8 | 5 | 5 | 5 | 3 | 13 | 12 | 10
nmol/L | 326 [241 to 442] | 680 [502 to 922] | 918 [653 to 1290] | 1250 [874 to 1790] | 373 [235 to 592] | 817 [514 to 1300] | 1300 [819 to 2060] | 1330 [837 to 2120] | 644 [522 to 796] | 1280 [1030 to 1600] | 1290 [1010 to 1630]

13. Secondary Outcome: Part 2: Tmax of MK-8189
Description: Tmax was determined for participants in Part 2 panels who received MK-8189.
Time Frame: Days 1, 4, 7, 10, and 13: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2, Panel D: MK-8189 8 mg | Part 2, Panel D: MK-8189 16 mg | Part 2, Panel D: MK-8189 24 mg | Part 2, Panel D: MK-8189 24 mg Day 13 | Part 2, Panel F: MK-8189 8 mg | Part 2, Panel F: MK-8189 16 mg | Part 2, Panel F: MK-8189 24 mg | Part 2, Panel F: MK-8189 24 mg Day 13 | Part 2, Panel G: MK-8189 16 mg | Part 2, Panel G: MK-8189 24 mg | Part 2, Panel G: MK-8189 24 mg Day 10
Number analyzed (Participants) | 12 | 12 | 9 | 8 | 5 | 5 | 5 | 3 | 13 | 10 | 10
Hours | 23.90 [10.00 to 24.00] | 14.00 [0.00 to 23.97] | 16.02 [0.00 to 24.00] | 10.08 [0.00 to 24.00] | 16.10 [16.00 to 23.95] | 16.07 [11.92 to 23.92] | 15.97 [11.92 to 16.00] | 16.00 [0.00 to 16.00] | 16.17 [10.00 to 23.98] | 11.99 [0.00 to 16.00] | 15.88 [0.00 to 23.95]

14. Secondary Outcome: Part 2: CL/F of MK-8189
Description: CL/F was determined for participants in Part 2 panels who received MK-8189.
Time Frame: Days 10 and 13: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Groups:
- Part 2, Panel D: MK-8189 24 mg: The PK of MK-8189 24 mg was assessed on Day 13 in Panel D.
- Part 2, Panel F: MK-8189 24 mg: The PK of MK-8189 24 mg was assessed on Day 13 in Panel F.
- Part 2, Panel G: MK-8189 24 mg: The PK of MK-8189 24 mg was assessed on Day 10 in Panel G.
Arm/Group | Part 2, Panel D: MK-8189 24 mg | Part 2, Panel F: MK-8189 24 mg | Part 2, Panel G: MK-8189 24 mg
Number analyzed (Participants) | 8 | 3 | 10
L/hr | 2.67 (28.5) | 2.18 (57.3) | 2.34 (29.8)

15. Secondary Outcome: Part 2: t½ of MK-8189
Description: t½ was determined for participants in Part 2 panels who received MK-8189.
Time Frame: Days 10 and 13: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2, Panel D: MK-8189 24 mg | Part 2, Panel F: MK-8189 24 mg | Part 2, Panel G: MK-8189 24 mg
Number analyzed (Participants) | 6 | 3 | 10
Hours | 13.98 (51.0) | 8.90 (33.4) | 9.99 (27.4)

16. Secondary Outcome: Part 2: Vd/F of MK-8189
Description: Vd/F was determined for participants in Part 2 panels who received MK-8189.
Time Frame: Days 10 and 13: Predose and 2, 6, 8, 10, 12, 16, and 24 hours postdose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 2, Panel D: MK-8189 24 mg Day 13 | Part 2, Panel F: MK-8189 24 mg | Part 2, Panel G: MK-8189 24 mg
Number analyzed (Participants) | 6 | 3 | 10
Liters | 55.23 (52.3) | 27.94 (57.2) | 32.91 (26.8)

ADVERSE EVENTS:
Time Frame: Up to approximately 27 days
Description: All randomized participants received ≥1 dose of study therapy and are included in all cause mortality and safety assessment.
Groups:
- MK-8189 8 mg: All participants who received MK-8189 8 mg are included.
- MK-8189 16 mg: All participants who received MK-8189 16 mg are included.
- MK-8189 24 mg: All participants who received MK-8189 24 mg are included.
- Placebo: All participants who received placebo are included.
- MK-8189 Total: All participants in Parts 1 and 2 who received any dose of MK-8189 are included.
- Total Participants: All study participants in Parts 1 and 2 are included.
Arm/Group | MK-8189 8 mg | MK-8189 16 mg | MK-8189 24 mg | Placebo | MK-8189 Total | Total Participants
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/36 | 0/45 | 0/13 | 0/50 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/36 | 0/45 | 0/13 | 0/50 | 0/63
Other Adverse Events (participants affected / at risk) | 5/17 | 19/36 | 26/45 | 6/13 | 36/50 | 42/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8189 8 mg (N=17) | MK-8189 16 mg (N=36) | MK-8189 24 mg (N=45) | Placebo (N=13) | MK-8189 Total (N=50) | Total Participants (N=63)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 3 (4) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 3 (3)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 5 (6) | 5 (6)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (3)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 5 (5) | 6 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dystonia (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 3 (4) | 4 (6)
Hypertonia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 4 (4)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Oromandibular dystonia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 7 (7) | 3 (3) | 1 (1) | 11 (11) | 12 (12)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Apathy (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Hallucination, tactile (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (2)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypnagogic hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 2 (3)
Nightmare (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (2)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT04506905/Prot_SAP_000.pdf